CLINICAL TRIAL: NCT04848181
Title: The Effect of Short Term Use of Finasteride Versus Cyproterone Acetate on Perioperative Blood Loss With Mono Polar Transurethral Resection of Prostate
Brief Title: The Effect of Pre-operative Use of Finasteride Versus Cyproterone Acetate on Blood Loss With Transurethral Resection of Prostate
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Shabieb Ahmed, shabieb ahmed ( assistant professor - urology department - Benha University), Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: benign prostatic hyperplasia
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Cyproterone Acetate; Finasteride

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- cyproterone acetate (Active Comparator): 20 patients received cyproterone acetate 50 mg twice per day for two weeks before TURP
  Interventions: Drug: cyproterone acetate
- finasteride group (Active Comparator): 20 patients received finasteride 5 mg once per day for two weeks before TURP
  Interventions: Drug: finasteride
- control group (Placebo Comparator): 20 patients received no treatment before TURP
  Interventions: Drug: no treatment received

INTERVENTIONS:
Drug: cyproterone acetate — two weeks Cyproterone acetate administration before TURP
  Arms: cyproterone acetate
Drug: finasteride — two weeks finasteride administration before TURP
  Arms: finasteride group
Drug: no treatment received — no treatment received before TURP
  Arms: control group

SUMMARY:
Perioperative bleeding is the most common complication related to transurethral resection of prostate, the aim of the study is to compare the effect of pre-operative use of finasteride versus Cyproterone acetate on blood loss with mono polar TURP

DETAILED DESCRIPTION:
This prospective randomized controlled study to compare the effect of pre-operative use of finasteride versus Cyproterone acetate on blood loss with mono polar TURP

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign prostatic hyperplasia with prostate size (60-100) grams
* Lower urinary tract symptoms (LUTS) not responding to medical treatment
* Recurrent prostatic bleeding
* Recurrent acute urinary retention
* Chronic urinary retention

Exclusion Criteria:

* Patients with coagulation disorders
* Previous prostatic surgery
* Previous finasteride administration
* Bladder pathology (urinary bladder stones - bladder mass)
* Suspected or proved cancer prostate
* Hepatic or renal impairment
* Patients unfit for operation eg. Decompensated heart failure, poor chest condition

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
post operative Hb | 24 hour post operative
  measuring serum haemoglobin level at first post operative
post operative Hcv | 24 hour post operative
  measuring serum haematocrit value at first post operative
operative duration | immediately after surgery
  assessment of the duration of the operation
microvascular density(MVD) | 2 weeks after drug intake
  assesment of MVD of the prostate by histological examination using high power field microscope
intraoperative blood loss | immediately after surgery
  assessment of intraoperative blood loss during TURP

CONTACTS AND LOCATIONS:
Overall Officials: shabieb ahmed, Ph.D, Study Director — faculty of medicine, Benha university; abdallah fathy, Ph.D, Study Director — faculty of medicine, Benha university; mohamed hefnawy, Ph.D, Study Chair — faculty of medicine, Benha university; adel al falah, Ph.D, Principal Investigator — faculty of medicine, Benha university
Locations (1):
- Benha University, Banhā, Qalyubia Governorate, Egypt

REFERENCES:
- [Background] Treharne C, Crowe L, Booth D, Ihara Z. Economic Value of the Transurethral Resection in Saline System for Treatment of Benign Prostatic Hyperplasia in England and Wales: Systematic Review, Meta-analysis, and Cost-Consequence Model. Eur Urol Focus. 2018 Mar;4(2):270-279. doi: 10.1016/j.euf.2016.03.002. Epub 2016 Mar 23. PMID 28753756
- [Background] Yang TY, Chen M, Lin WR, Li CY, Tsai WK, Chiu AW, Ko MC. Preoperative treatment with 5alpha-reductase inhibitors and the risk of hemorrhagic events in patients undergoing transurethral resection of the prostate - A population-based cohort study. Clinics (Sao Paulo). 2018 Mar 12;73:e264. doi: 10.6061/clinics/2018/e264. PMID 29538495
- [Background] Khwaja MA, Nawaz G, Muhammad S, Jamil MI, Faisal M, Akhter S. The Effect of Two Weeks Preoperative Finasteride Therapy in Reducing Prostate Vascularity. J Coll Physicians Surg Pak. 2016 Mar;26(3):213-5. PMID 26975954
- [Background] Tian HL, Zhao CX, Wu HY, Xu ZX, Wei LS, Zhao RT, Jin DL. Finasteride reduces microvessel density and expression of vascular endothelial growth factor in renal tissue of diabetic rats. Am J Med Sci. 2015 Jun;349(6):516-20. doi: 10.1097/MAJ.0000000000000451. PMID 25789687
- See also: Transurethral Resection of Prostate is Still the Gold Standard for Small to Moderate Sized Prostates — https://www.journal-ina.com/text.asp?2016/3/2/68/181223